CLINICAL TRIAL: NCT03337815
Title: A 24-Week, Multicenter ,Double Blind, Randomized Study to Determine the Effects and Security of Tripterygium Wilfordii Treating Rheumatoid Arthritis and Establish A Prediction Model
Brief Title: A Specification Clinical Application Research of Tripterygium Wilfordii Treating Rheumatoid Arthritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Quan Jiang, director, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Z161100000516020-1
Record Dates: First submitted 2017-10-22; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of MTX and TwHF placebo (Active Comparator): Patients were treated with Methotrexate (MTX) and Tripterygium wilfordii Hook F（TwHF）placebo.
  Interventions: Drug: Treatment of MTX and TwHF placebo
- Treatment of TwHF and MTX placebo (Experimental): Patients were treated with Tripterygium wilfordii Hook F（TwHF）and Methotrexate (MTX) placebo.
  Interventions: Drug: Treatment of TwHF and MTX placebo

INTERVENTIONS:
Drug: Treatment of MTX and TwHF placebo — Methotrexate: 10-15mg per week according to patient's weight, oral, for 24 weeks.Tripterygium wilfordii Hook F（TwHF）placebo：20mg,3 times a day, oral, for 24 weeks.
  Arms: Treatment of MTX and TwHF placebo
Drug: Treatment of TwHF and MTX placebo — Tripterygium wilfordii Hook F（TwHF)：20mg,3 times a day, oral, for 24 weeks.Methotrexate (MTX)placebo: 10-15mg per week according to patient's weight, oral, for 24 weeks.
  Arms: Treatment of TwHF and MTX placebo

SUMMARY:
Rheumatoid Arthritis (RA) is an autoimmune disease that results in a chronic inflammatory disorder that may affect many synovial joints, and may cause serious disability. It has been confirmed that Tripterygium Wilfordii has effects of anti-inflammatory, immunosuppressive and cartilage protection. This is a multicenter ,double Blind, randomized study to evaluated the efficacy and safety of Tripterygium Wilfordii in treating of patients with rheumatoid arthritis (RA) and establish a prediction model for Tripterygium Wilfordii response of rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
Two arms were included in this study. Active Comparator: Patients were treated with Methotrexate (MTX)and Tripterygium wilfordii Hook F（TwHF）placebo.Experimental:Patients were treated with Methotrexate (MTX) placebo and Tripterygium wilfordii Hook F（TwHF)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with rheumatoid arthritis as determined by the 1987 or 2010 ACR classification criteria;
* No male or female fertility requirements, or around menopause women;
* Patients with mild-to-moderate activity, 2.6 < DAS28≤5.1;
* No serious system involved, such as severe pericardial effusion, interstitial lung disease, renal tubular acidosis, atrophic gastritis, autoimmune liver disease, etc;
* Within a month before the selected participants did not attend any drugs

Exclusion Criteria:

* Patients with cancer or other malignant disease such as cardiovascular, hematopoietic, liver and kidney disease, and psychopath
* Active or chronic infection, including HIV, hepatitis C virus, hepatitis B virus, tuberculosis
* Previous treated with tripterygii, glucocorticoid or biologic disease-modifying antirheumatic drug (DMARD) in 3 months.
* Previous treated with Tripterygium Wilfordii or MTX
* Patients with retinopathy.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2017-10-28 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
The change in Disease Activity Score (DAS28) | 0 weeks, 4 weeks，12 weeks, 24 weeks,52 weeks
  Disease Activity Score for 28-joint counts was based on the erythrocyte sedimentation rate(ESR) (DAS28-4[ESR])

SECONDARY OUTCOMES:
The proportion of patients achieving ACR20/50/70 | 0 weeks, 4 weeks，12 weeks, 24 weeks
  ACR20/50/70 is referred to American College of Rheumatology Criteria
The change in Health Assessment Questionnaire (HAQ) score | 0 weeks, 4 weeks，12 weeks, 24 weeks,52 weeks
  HAQ scores ranges from 0 to 3, with higher scores indicating greater disability
The change in Sharp scoring system of van der Heijde(Sharp) score | 0 week,24 weeks,52 weeks
  The change in Sharp score from baseline to week 24 and 52.According to the revised Sharp scoring system of van der Heijde, the joint gap score was scored in 30 regions of the hands (score range 0-120 points), and the bone erosion score was conducted in 32 areas (score range 0-160).The higher the score, the more serious the joint destruction.
The number of adverse events | 24 weeks
  The number of adverse events that are related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Quan, MD, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No